CLINICAL TRIAL: NCT02843087
Title: The Breastfeeding and Early Child Health (BEACH) Study
Brief Title: Pediatric Obesity and the Infant Microbiome (BEACH)
Acronym: BEACH
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201601034; OCR16157 (Other: University of Florida); 1K01DK115632-01A1 (NIH)
Record Dates: First submitted 2016-07-07; First posted 2016-07-25 (Estimated); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Pediatric Obesity
Keywords: Breastfeeding; Microbiome; BEACH; Human milk; Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Non- invasive biospecimens include stool, saliva, blood, urine, human milk, and vaginal swab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- NW vaginal deliveries: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center. Infant body composition is the primary outcome and will be monitored via anthropometry.
- NW C-section deliveries: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center. Infant body composition is the primary outcome and will be monitored via anthropometry.
- Ob vaginal deliveries: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center. Infant body composition is the primary outcome and will be monitored via anthropometry.
- Ob C-section deliveries: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center. Infant body composition is the primary outcome and will be monitored via anthropometry.
- GDM vaginal deliveries: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center. Infant body composition is the primary outcome and will be monitored via anthropometry.
- GDM C-section deliveries: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center. Infant body composition is the primary outcome and will be monitored via anthropometry.
- T2D vaginal deliveries: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center. Infant body composition is the primary outcome and will be monitored via anthropometry.
- T2D C-section deliveries: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center. Infant body composition is the primary outcome and will be monitored via anthropometry.
- T1D vaginal deliveries: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center. Infant body composition is the primary outcome and will be monitored via anthropometry.
- T1D C-section deliveries: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center. Infant body composition is the primary outcome and will be monitored via anthropometry.

SUMMARY:
The impact of breastfeeding on the infant microbiome in vaginally and Cesarean delivered offspring from obese and normal weight mothers.

DETAILED DESCRIPTION:
Design: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center.

Infant body composition is the primary outcome and will be monitored via anthropometry. Follow-up data points will be collected from electronic health records (EHR) and include but are not limited to wellness visits by 1 month, 2 months, 4 months, 6 months, 9 months, 12 months, 15 months, 18 months, 2 years, 2 ½ years, 3 years, and each year after that until 17.9 years. Planned data analysis includes linear regression using the R statistical program. The primary data analysis will test maternal health status and human milk bioactive components for associations with the infant microbiome and pediatric outcomes collected by clinical visits and EHR.

The study team will recruit equal samples of pregnant mothers in each the following groups (n=50 in each group; 1800 total participants): 1) NW vaginal deliveries; 2) NW C-section deliveries; 3) Ob vaginal deliveries 4) Ob C-section deliveries; 5) GDM vaginal deliveries; 6) GDM C-section deliveries; 7) T2D vaginal deliveries; 8) T2D C-section deliveries; 9) T1D vaginal deliveries; 10) T1D C-section deliveries.

Stool, saliva, and vaginal swab samples collected from participants may be used for animal studies whereby germ-free mice are inoculated with stool samples to evaluate a causal role of the microbiome in clinically relevant phenotypes (i.e. pediatric obesity).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 45 years of age.
* Pre-pregnancy BMI is greater than 30 kg/m2
* Pre-pregnancy BMI is less than 25 kg/m2
* At risk for gestational diabetes
* Pregnant and have Type 1 diabetes (T1D)
* Pregnant and have Type 2 diabetes (T2D)
* pregnant and within the 3rd trimester (34-36 weeks of gestation)-You plan to deliver in the Greater Gainesville area
* Plan to deliver via vaginal or cesarean section
* Plan to exclusively breastfeed your infant for at least 2 months
* Child will receive their pediatric care through UFHealth

Exclusion Criteria:

* Smoking
* Pre-eclampsia
* History of pre-term delivery (<35 weeks)
* Only one breast capable of lactation and milk production inadequate
* Age <18 yrs, >45 yrs
* Any maternal antibiotics in the last 2 weeks during delivery
* Any alcohol consumption
* Drug use

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal weight (NW; pre-pregnant BMI <25.0 kg/m2), obese (Ob; pre-pregnant BMI >30.0 kg/m2), gestational diabetes (GDM), Type 2 diabetes (T2D), and Type 1 diabetes mothers during the 3rd trimester (34-36 weeks) of pregnancy that will be followed -along with their respective offspring- through the first 12 months of life will be recruited from the University of Florida (UF) Health Shands Hospital. Stool, saliva, blood, vaginal swab, human milk, urine, body composition and clinical variables will be collected from mother and infant at 34-36 weeks of gestation (mom only), 2-weeks, 2-months, and 1-year at the UF Clinical Research Center.
  The following groups (n=50 in each group; 1800 total participants): 1) NW vaginal deliveries; 2) NW C-section deliveries; 3) Ob vaginal deliveries 4) Ob C-section deliveries; 5) GDM vaginal deliveries; 6) GDM C-section deliveries; 7) T2D vaginal deliveries; 8) T2D C-section deliveries; 9) T1D vaginal deliveries; 10) T1D C-section deliveries.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Measure bioactive compounds in human milk (HM) via Enzyme-linked immunosorbent assay (ELISA) | 1 year
Quantify the infant intestinal gene expression profile in stool by real-time polymerase chain reaction (PCR) | 1 year
Measure the infant intestinal gene expression profile in stool via whole genome sequencing (WGS). | 1 year

SECONDARY OUTCOMES:
Measure Body Mass Index (BMI) in kg/m^2 via the Body Bod instrument. | 1 year
Measure weight in kilograms by using a body weight scale. | 1 year
Measure height in meters via stadiometer. | 1 year

OTHER OUTCOMES:
Measure infant body composition by using anthropometry. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Lemas, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH Data Sharing Policy of award 1U24DK097193, all data generated by Southeast Center for Integrated Metabolomics (SECIM), along with the corresponding metadata, will be deposited into the NIH Metabolomics Data Repository and Coordinating Center (DRCC) as soon as all quality control steps are completed. Data will be embargoed for one year and, after the expiration of the embargo, made visible to the scientific community regardless of publication status for the data.